CLINICAL TRIAL: NCT05644249
Title: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) and Systemic Chemotherapy as a First-line Treatment for Gastric Cancer Peritoneal Metastases: Open-label, Single-arm, Multi-center Feasibility Study
Brief Title: PIPAC and FOLFOX for Gastric Cancer Peritoneal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Vilnius University Hospital Santaros Klinikos (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Martynas Luksta, Abdominal surgeon, Vilnius University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1
Record Dates: First submitted 2022-09-29; First posted 2022-12-09 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
Keywords: Gastric cancer; Peritoneal carcinomatosis; PIPAC; FOLFOX; Bidirectional
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental treatment (Experimental): Each patient will be scheduled for 3 courses of combined treatment: in total 3 PIPAC with cisplatin 10.5 mg/m2 and doxorubicin 2.1 mg/m2 and 6 cycles of FOLFOX systemic chemotherapy.
  Interventions: Drug: Combined Doxorubicin and Cisplatin Pressurized IntraPeritoneal Aerosol Chemotherapy With Systemic FOLFOX chemotherapy

INTERVENTIONS:
Drug: Combined Doxorubicin and Cisplatin Pressurized IntraPeritoneal Aerosol Chemotherapy With Systemic FOLFOX chemotherapy — Each course of combined treatment will start with PIPAC (a pressurized aerosol containing cisplatin 10.5 mg/m2 and doxorubicin 2.1 mg/m2 diluted in NaCl 0.9% applied through the nebulizer inside the abdominal cavity during laparoscopy). Fourteen days afterward 2 cycles of systemic FOLFOX chemotherapy will be applied within 28 days. The interval between combined treatment courses will be 14 days.
  Other Names: PIPAC

SUMMARY:
Peritoneum is among the most common sites of metastases in gastric cancer. Systemic chemotherapy is the current standard for peritoneal carcinomatosis (PC), although, the treatment results remain extremely poor. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a modern treatment modality for PC, that 1) optimize the drug distribution by applying an aerosol rather than a liquid solution; and 2) apply increased intraperitoneal hydrostatic pressure to increase drug penetration to the target. Despite some encouraging preliminary results for PIPAC efficacy, it is still an investigational treatment. Furthermore, only very limited data exist for bidirectional treatment, which includes a combination of systemic chemotherapy and PIPAC. Thus, this study will investigate the feasibility of PIPAC and systemic chemotherapy combination for gastric cancer patients with peritoneal metastases.

DETAILED DESCRIPTION:
This open-label, single-arm feasibility study will be conducted at two major gastrointestinal cancer treatment centers in Lithuania and will include 37 participants. Gastric cancer patients diagnosed with a synchronous or metachronous peritoneal carcinomatosis based on a clinical, radiological, cytological, and histological examination will be considered for enrollment. Thirty-seven patients willing to participate and meeting the enrollment criteria will be scheduled for the experimental treatment. Three cycles of 1st line palliative systemic chemotherapy will be administered every 28 days and PIPAC with cisplatin 10,5 mg/m2 and doxorubicin 2,1 mg/m2 will be utilized 14 days after each of the systemic chemotherapy cycles. After the 3rd PIPAC procedure patients will be re-assessed and discussed at multidisciplinary team meetings. In case of downstaging patients will be considered for radical gastrectomy±cytoreductive surgery; others for further systemic therapy. All patients will be followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically verified gastric adenocarcinoma (HER2 negative) with peritoneal carcinomatosis;
2. Age≥18;
3. ECOG≤1;
4. Patient willing to participate;
5. Patient is the candidate for 1st line FOLFOX palliative systemic chemotherapy.

Exclusion Criteria:

1. Extra-abdominal metastases;
2. Siewert I type gastroesophageal junction cancer;
3. Mechanical bowel obstruction;
4. Allergy to study drugs;
5. History of previous intraperitoneal chemotherapy;
6. Pregnancy of refusal for birth-control at least 6 months post-study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Objective tumor response according to RECIST v 1.1 after second PIPAC | Day 7 after second PIPAC procedure (an average of 8 weeks after start of the study)
  Objective tumor response according to RECIST v 1.1 in CT scan performed 1 week after second PIPAC procedure

SECONDARY OUTCOMES:
Objective tumor response according to RECIST v 1.1 | Day 7 after third PIPAC procedure (an average of 15 weeks after start of the study)
  Objective tumor response according to RECIST v 1.1 in CT scan performed 1 week after third PIPAC procedure
Compliance to treatment | Through study completion, an average of 28 months
  Proportion of patients able to receive all anticipated treatment (3 PIPACs and 6 cycles of FOLFOX)
Postoperative complication assessed by Clavien-Dindo score | Through study completion, an average of 28 months
  The number of patients with postoperative complications, defined and graded according to Clavien-Dindo classification
Peritoneal carcinomatosis index and histological regression according to peritoneal regression grading score (PRGS). | Through study completion, an average of 28 months
  A pathologist blinded to clinical outcomes will evaluate histological tumor response using the Peritoneal Regression Grading Score (PRGS): 1-Complete regression without cancer cells; 2-higher response with prevalence of regressive phenomena and only a few residual cancer cells - PRGS; 3-minor response with prevalence of residual cancer cells and poor regressive phenomena; 4-no response to therapy without regressive phenomena.
  A patient will be considered a responder if any reduction in the PRGS during subsequent biopsies will be recorded.
Ascites volume | Through study completion, an average of 28 months
  The volume of ascites recorded at every PIPAC procedure.
Tumor markers | Through study completion, an average of 28 months
  Ca19-9, carcinoembryonic antigen (CEA), Ca72-4 plasma levels measured at different time points.
Quality of life by EORTC questionnaires | Through study completion, an average of 28 months
  Quality of life by EORTC questionnaires measured at different time points.
Overall survival | From treatment start to death, assessed up to 24 months
  Time from start of the treatment to death
Progression-free survival | From treatment start to death, assessed up to 24 months
  Time from start of the treatment to progression of the disease
Adverse events of chemotherapy drugs | Through study completion, an average of 28 months
  The number of patients with toxicity according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0 during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Skaiste Tulyte, MD, Principal Investigator — Vilnius University Hospital Santaros Klinikos
Locations (2):
- Lithuania (2):
  - Nationa Cancer Institute, Vilnius, Vilniaus
  - Vilnius University hospital Santaros Klinikos, Vilnius, Vilniaus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luksta M, Bausys A, Bickaite K, Rackauskas R, Paskonis M, Luksaite-Lukste R, Ranceva A, Stulpinas R, Brasiuniene B, Baltruskeviciene E, Lachej N, Sabaliauskaite R, Bausys R, Tulyte S, Strupas K. Pressurized intraperitoneal aerosol chemotherapy (PIPAC) with cisplatin and doxorubicin in combination with FOLFOX chemotherapy as a first-line treatment for gastric cancer patients with peritoneal metastases: single-arm phase II study. BMC Cancer. 2023 Oct 25;23(1):1032. doi: 10.1186/s12885-023-11549-z. PMID 37875869